CLINICAL TRIAL: NCT03889054
Title: Effect of a Joint Program of Health Education and Respiratory Rehabilitation on the Health-related Quality of Life of Patients With Chronic Obstructive Pulmonary Disease and History of Exacerbation
Brief Title: Effect of Education and Respiratory Rehabilitation on Quality of Life in COPD Patients
Acronym: EDUEPOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI-3534
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Randomized and parallel clinical trial of 66 patients (33 with health education associated with respiratory rehabilitation and 33 only with respiratory rehabilitation). There will be a follow-up of 6 months and 4 visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Current clinical management
- Structured health education program (Active Comparator): Patient will be referred to a specific consultation to carry out this intervention.
  Interventions: Behavioral: Education program

INTERVENTIONS:
Behavioral: Education program — The education sessions will be given in 3 opportunities (15-30, 45 and at 90 days from diagnosis of the exacerbation) and it will be individualized. The program will include measures of self-care and self-management recommended in patients with COPD:
  1. Plan of action in an exacerbation.
  2. Education related to COPD.
  3. Information on pharmacological medication.
  4. Management of the exacerbation.
  5. Management of stress and / or anxiety.
  6. Nutritional recommendations.
  7. Physical exercise recommendations.
  8. Healthy lifestyle recommendations. The first session will last 90 minutes and will be explain according to the contents of the manual "Controlling COPD". A presentation designed for this purpose will be displayed and this manual will be provided to patients to carry out their reading at home. The second and third sessions will last 15 minutes and the purpose will be to resolve doubts.
  Other Names: Behavioral management
  Arms: Structured health education program

SUMMARY:
In patients with COPD and a history of recent exacerbation, to compare the quality of life after completing a joint program of health education and respiratory rehabilitation with those patients who only receive respiratory rehabilitation. To compare lung function, the distance traveled in the 6-minute walk test and in the test of the shuttle between both groups. Also, to compare between both groups adherence to inhaled treatment, physical activity, and emotional condition. Finally, to compare the number of visits to emergencies and hospitalizations, and on the other hand, the number of mild, moderate and severe exacerbations between both groups

DETAILED DESCRIPTION:
In this trial we selected COPD patients with a history of recent exacerbation to be submitted to a respiratory rehabilitation program with or without a individualized program of health education. We try to demonstrate a better improvement in the quality of life after completing a joint program of health education and respiratory rehabilitation in this patients than those one who only receive respiratory rehabilitation. We also want to demonstrate an improvement in lung function, the distance travelled in the 6-minute walk test and in the test of the shuttle, the adherence to inhaled treatment, the physical activity, the emotional condition, the number of visits to emergencies and hospitalizations and the number of mild, moderate and severe exacerbations between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age over 30 years.
* COPD diagnosis according to GesEPOC criteria (FEV 1 / FVC greater 0.7).
* Smoker or ex-smoker with a cumulative consumption of more than 10 packages per year.
* Exacerbation of COPD diagnosed in the last 15 days.

Exclusion Criteria:

* Impossibility of obtaining informed consent.
* Osteoarticular, neuromuscular or cognitive limitation.
* Diagnosis of active neoplastic disease, except epidermoid carcinoma of skin.
* Patient with limitation or difficulty to go to the rehabilitation unit to complete the training program.
* Participation in another study / trial in the previous 6 months.
* Have participated in a respiratory rehabilitation program the previous year (12 previous months).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life after 6 months of education | Six months
  To compare the quality of life related to health measured by the Saint George respiratory questionnaire after 6 months between patients who received health education and those who did not receive it.
Quality of life after 6 months of education | Six months
  To compare health relate quality of life measured by the EuroQoL questionnaire, after 6 months between patients who received health education and those who did not receive it.
Quality of life after 6 months of education | Six months
  To compare health relate quality of life measured by COPD Assessment Test (CAT) after 6 months between patients who received health education and those who did not receive it.

SECONDARY OUTCOMES:
Pulmonary function after 6 months of education | Six months
  To compare pulmonary function measured by spirometry after 6 months between patients who received health education and those who did not receive it.
Distance traveled in the 6-minute walk test and in the shuttle walking test after 6 months of education | Six months
  To compare the distance traveled in the 6-minute walk test and in the shuttle walking test after 6 months between patients who received health education and those who did not receive it.
Adherence to inhaled treatment after 6 months of education | Six months
  To compare adherence to inhaled treatment after 6 months between patients who received health education and those who did not receive it.
Physical activity of patients after 6 months of education | Six months
  To compare the physical activity of patients measured by International Physical Activity Questionnaire (IPAQ) after 6 months between patients who received health education and those who did not receive it.
Physical activity of patients after 6 months of education | Six months
  To compare the physical activity of patients measured by an accelerometer after 6 months between patients who received health education and those who did not receive it.
Emotional state of patients after 6 months of education | Six months
  To compare the emotional state of patients measured by Hospital Anxiety and Depression Scale (HADS) after 6 months between patients who received health education and those who did not receive it.
Number of visits to the emergency department, number of hospital admissions and days of hospital admission of patients after 6 months of education | Six months
  To compare the number of visits to the emergency department, the number of hospital admissions and the days of hospital admission after 6 months between patients who received health education and those who did not receive it.
Number of mild, moderate and severe exacerbations of patients after 6 months of education | Six months
  To compare the number of mild, moderate and severe exacerbations after 6 months between patients who received health education and those who did not receive it.

IPD SHARING:
Plan to Share IPD: No